CLINICAL TRIAL: NCT03903055
Title: Study on Improving Clinical Diagnosis Classification and Prognosis Evaluation Criteria and Precise Early Intervention Treatment of High-risk MDS Patients Based on RNA-seq Technology
Brief Title: Study on High-risk MDS Patients Based on RNA-seq Technology
Acronym: MDS&RNA-seq
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Provincial Hospital of TCM (Other)
Responsible Party: Principal Investigator, Shengyun Lin, Clinical Professor, Zhejiang Provincial Hospital of TCM
Other Study IDs: 2018C03G2120113
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: MDS
Keywords: MDS; RNA-seq

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MDS group — patients diagnosed as MDS with high risk，aged 18-80，men/wemen

SUMMARY:
MDS is a group of malignant cloned blood diseases that originated from hematopoietic stem cells(HSC) or CD34 + progenitor cells and are still incurable. Its main characteristics are the increase of primitive cells in the bone marrow accompanied by a series or multiple developmental abnormalities(pathological hematopoiesis), the reduction of peripheral blood cells, the high risk of conversion to acute myeloid leukemia(AML), and once converted to leukemia, the treatment prognosis is very poor.The bone marrow cells of MDS patients were deeply sequenced by RNA-Seq method. Through differential gene expression analysis, different genes related to the onset and evolution of MDS were selected and their expression levels were analyzed in different subtype MDS patients. To study its significance in clinical classification, prognosis assessment and early intervention treatment, establish a new standard for clinical classification and prognosis evaluation based on genomic classification, clarify early intervention or precise treatment schemes, and significantly prolong the survival of patients, Improving the quality of life.

DETAILED DESCRIPTION:
(1) Study population(included in the standard): 120 patients(aged 16 to 80 years) who met the MDS diagnostic criteria in the hematology department and outpatient clinics of the four cooperative hospitals after June 2019. The diagnostic criteria refer to the WHO diagnosis of the 2016 MDS. New classification; The prognosis score was based on the 2012 MDS revised IPSS-R prognostic integral system.In control group, 5 patients with initial acute myeloid leukemia(AML-M2a) and 5 healthy human bone marrow donation volunteers. Understand the purpose of this study and sign an informed consent form.

2) Clinical information collection: medical history collection of selected patients, Routine clinical tests(including peripheral blood count, serum ferritin, VitB12, folic acid, EPO levels, bone marrow smears and bone marrow biopsies, bone marrow flow cytometry, bone marrow cytogenetics, etc.) and follow-up and efficacy observations, The clinical indicators, efficacy and prognosis of the patient and the possible related genes detected were systematically analyzed.

(3) Research methods: The bone marrow specimens collected will be extracted according to the RAN-seq operating process, and the total RNA, quality test, and cDNA library of each sample cell will be extracted, 30 Million reads per sample, and Ilumina X10 PE150 will be sequenced, sequencing depth 9G clear Data. After the sequencing data is tested and passed, the original sequencing data is pre-processed: the raw data of the sequencing machine is qualitatively controlled, the sequencing fragments with the sequencing connector are removed, and the low-quality, fuzzy N bases, riboomeRNA are removed. Sequencing fragments with a length of less than 20, etc.; Transcription of sequencing data: genomic alignment of preprocessed reads and post-comparison quality control.

Gene Expression Level Analysis: Gene Expression Level Quantification, Gene Expression Level Distribution, Biological Duplication Correlation Analysis, Intersample Level Clustering and PCA Analysis.

Differential Expression Gene Analysis:

The GO enrichment and signal pathway enrichment of different genes were analyzed, and the genes specifically raised or decreased between normal samples, AML samples, and MDS patient samples(including various MDS subtypes) were compared. Prediction of molecular level events associated with these differential gene changes(signal pathway activation or inhibition), and search for differential genes that can represent disease processes.

(4) Data management and statistics: All clinical information data are collected and entered into the computer. All data are entered using the database established by the Clinical Evaluation and Analysis Center of the unit. Data processing statisticians finally further fully verify and check the completeness and accuracy of data before data entry. Data entry and management by the person responsible for the establishment of a dedicated database, data entry and management should be entered and proofread by two data managers. After completion, SPSS 19.0 for Windows statistics software package is used for statistical processing.

After the completion of clinical information data statistics and sequencing analysis results, the computer's "in-depth learning" function was used to complete the establishment of two "standards" and one "scheme" using analysis tools such as rMATS and SURVIV.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet MDS diagnostic criteria with high risk of IPSS-R

Exclusion Criteria:

with no MDS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the population of MDS patients were from the five centers who were visiting the doctor
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
RNA-seq | 2021-2022
  use questionnaire to research whether the target mutation gene combination analyzed by transcription group was consistent with clinical cell morphological diagnosis and disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: lin s yun, doctor, Study Chair — zjhtcm
Locations (1):
- ZJHTCM, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided